CLINICAL TRIAL: NCT02363816
Title: Beta-carotene and Oxidative Stress in Pediatric Second Generation Antipsychotic Use
Status: Withdrawn | Type: Observational
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Kyle Burghardt, Assistant Professor, Wayne State University
Other Study IDs: PEDSGAWSU
Record Dates: First submitted 2014-08-28; First posted 2015-02-16 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Pediatric Population on Second Generation Antipsychotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Weight gain, hypertension, high cholesterol and sugar abnormalities in childhood are strongly linked and predict the risk of further complications and early death in adulthood. The newer antipsychotics, called the second generation antipsychotics are commonly used to treat mood disorders in adult and pediatric populations. Their use has substantially increased (up to 5-fold) in the past 15 years in children due to their approved use by the Food and Drug Administration and higher acceptance in the general medical community. However, second generation antipsychotics are known to have very damaging side effects that cause children to gain substantial amounts of weight, have high cholesterol, high blood pressure and high sugar levels. Despite the known risks their use is still needed and may be contributing to the high rates of obesity-related diseases in childhood and ultimately shorter life-spans in adulthood. How second generation antipsychotics cause these side effects is still not well known. Preliminary evidence has identified a novel pathway that may be associated with second generation antipsychotic side effects. This pathway has not been studied, is involved in vitamin A metabolism and is called the beta-carotene pathway. Beta-carotene is an important part of our diet because it acts as an anti-oxidant (fights harmful oxidative stress in the body) and it produces the active form of vitamin A which is essential for several processes in our body. The investigator's work has identified a backup in this pathway which the investigators hypothesize is due to genetic variation of the enzymes found within this pathway.

The investigators hypothesize that genetic variation in the beta-carotene pathway is responsible for the side effects associated with second generation antipsychotics. The investigators want to complete a cross-sectional, pilot study in the pediatric population that will be used for future prospective, extramural applications.

The investigators propose two aims for this study:

Aim 1: Determine how second generation antipsychotics change beta-carotene metabolism. For this aim, the investigators hypothesize that high beta-carotene:retinoic acid ratios will be due to genetic varition in the beta-carotene pathway.

Aim 2: Define the relationship between beta-carotene metabolism, oxidative stress and second generation antipsychotic induced insulin resistance. For this aim the investigators hypothesize that low beta-carotene levels will be associated with high oxidative stress levels and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 10 to 17 years currently treated with one or more antipsychotics as determined by a physician
2. No changes in antipsychotic dosage for the past 6 weeks.

Exclusion Criteria:

1. Guardian or child unwilling or unable to participate.
2. A diagnosis of diabetes or dyslipidemia prior to starting an antipsychotic.
3. Abuse or dependence diagnoses

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric population treated with second generation antipsychotics
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
beta-carotene levels | measured during cross-sectional visit
  serum level reported in mcg/dL
retinoic acid levels | measured during cross-sectional visit
  serum level reported in nmol/L

SECONDARY OUTCOMES:
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | measured during cross-sectional visit
  Calculated by the following equation: [fasting insulin (pIU/mL) × fasting blood glucose (mmol/L)]/22.5
F2 Isoprostanes | measured during cross-sectional visit
  peripheral biomaker of oxidative stress determined by ELISA in pg/ml